CLINICAL TRIAL: NCT02741778
Title: Minimally Invasive Sweet Esophagectomy for Patients With Siewert Type II Adenocarcinoma of the Esophagogastric Junction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1501041143
Record Dates: First submitted 2015-11-02; First posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Adenocarcinoma
Keywords: Esophagogastric Junction; Adenocarcinoma; Cardia
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minimally invasive group (Other): In this group, all manipulations are finished by laparoscopy and thoracoscopy.
  1. Horizontal position, undergoing laparoscopy through 5-port method. The sequence: gastric mobilization, lymph nodes dissection(including paracardial nodes, left gastric nodes, and detecting splenic nodes and common hepatic nodes ), gastric tube making, and jejunostomy.
  2. Left lateral position, undergoing thoracoscopy through 3-port method. The sequence: mobilization of lower esophagus, lower paraesophagesl nodes and diaphragmatic nodes dissection, gastro-esophageal anastomosis by using CEEA.
  Interventions: Procedure: Minimally invasive group
- Open group (Other): Right lateral position, Traditional thoracotomy through the 7th intercostal incision. The sequence: mobilization of lower esophagus, lower paraesophagesl nodes and diaphragmatic nodes dissection.
  Then,oped the diaphragm,undergoing gastric mobilization, lymph nodes dissection(including paracardial nodes, left gastric nodes, and detecting splenic nodes and common hepatic nodes), gastric tube making, gastro-esophageal anastomosis by using CEEA. Nasointestinal tube is placed for feeding.
  Interventions: Procedure: Open group

INTERVENTIONS:
Procedure: Minimally invasive group — In this group, all manipulations are finished by laparoscopy and thoracoscopy.
  Arms: Minimally invasive group
Procedure: Open group — Right lateral position, Traditional thoracotomy through the 7th intercostal incision.
  Arms: Open group

SUMMARY:
Of the esophagogastric junction adenocarcinoma (AEG) is a 5 cm region of adenocarcinoma of the esophagus and stomach. Due to the special anatomical location, the biological behavior of esophageal cancer and gastric cancer are not the same. For the resection of esophageal gastric junction adenocarcinoma, the main treatment method for the treatment of surgical treatment.

For the type II type of esophageal gastric junction adenocarcinoma, the mainstream of the traditional surgical approach for the left chest to open the chest, for the lesions of the small type of esophageal gastric junction adenocarcinoma can be performed minimally invasive Ivor-Lewis esophageal resection.

There is no reasonable standard for treatment of type II type esophageal gastric junction adenocarcinoma. The investigators sum up the experience of the past in the minimally invasive resection of esophageal cancer, and combine domestic and foreign research results. Pioneered by laparoscopic mobilization of the stomach and dissection of the abdominal field lymph node + thoracoscopic (left thoracic approach) to free the esophagus and cleaning + mirror under the purse string forceps esophagogastric aortic arch anastomosis under lower mediastinal lymph node, corresponding to the operation is the traditional through left thoracotomy combined with open operation on diaphragm. Can achieve the same with the traditional surgical resection of the tumor, while taking into account the characteristics of minimally invasive surgery. This study intends to provide a minimally invasive surgical treatment of the chest laparoscopy combined with minimally invasive surgery and traditional thoracotomy. Comparison of different surgical methods for patients with the safety of surgery, oncology resection range, the incidence of short-term complications. The effect of different surgical methods on the survival rate and quality of life of the two groups were compared with the postoperative follow-up. The surgical treatment of esophageal carcinoma with a reasonable level of type II type of esophageal gastric junction adenocarcinoma is improved, and the surgical treatment of esophageal gastric junction adenocarcinoma is improved.

DETAILED DESCRIPTION:
Of the esophagogastric junction adenocarcinoma (AEG) is a 1 region of the 5 cm region in the esophageal gastric junction. Due to the special anatomical location, the biological behavior of esophageal cancer and gastric cancer are not the same. Because of its wide range of lesions, the majority of the Siewert classification system will be divided into three types: I type, CM type, CM 1-5, which is the 5 cm of the CM L, which is the traditional meaning of cardiac carcinoma. In the investigators country, the majority of patients with type II and III are 2,3,4. For the resection of esophageal gastric junction adenocarcinoma, the main treatment method for the treatment of surgical treatment. The high incidence of type II and type III AEG, type III patients more than the use of the abdominal approach to the proximal gastrectomy, more than by the Department of general surgery. In patients with lesions, the lymph node metastasis is also characterized by a bidirectional transfer of the lymph nodes and the peritoneal cavity with the lesion of the two boundary. In order to ensure that the upper cut edge of the esophagus and the dissection of the mediastinal lymph nodes, the domestic more by the Department of thoracic surgery. For the part of the patients, the traditional standard surgical approach to the left thoracic approach with open phrenoesophageal, partial resection of the stomach, aortic arch esophagogastric anastomosis + thoraco abdominal 2-field lymph node dissection dissection [5,6]. The minimally invasive surgery in the treatment of esophageal cancer and gastric cancer has been widely accepted by domestic and foreign counterparts. For I type AEG patients with type Ivor-Lewis and type III AEG patients are commonly used in the treatment of gastric cancer, and the corresponding minimally invasive surgery has a certain development [7,8]. And for type II AEG patients with relatively standard minimally invasive surgery, there is no unit carried out at home and abroad. Therefore, how to choose the minimally invasive method to complete this operation is more thorough. It has become a hot research topic in the domestic and foreign doctors. It has very important clinical significance and application prospect.

For the type II type of esophageal gastric junction adenocarcinoma, the mainstream of the traditional surgical method for the left chest approach to open the chest. The operation has the following disadvantages: 1) the integrity of the chest wall and diaphragm, the impact of the chest and abdomen of patients with large, close to the long-term life quality is greatly affected by the traditional surgery using the right side of the chest, abdominal lymph node dissection through the diaphragm to complete, and its complete abdominal approach to the poor. The foreign part of the center for smaller lesions of type II esophageal gastric junction adenocarcinoma underwent minimally invasive Ivor Lewis esophagectomy, but it exists the following drawbacks: 1) is not suitable for larger tumors; 2) gastric resection is not enough, the type of esophageal and gastric junction adenocarcinoma essence should be a special type of gastric carcinoma, proximal gastric resection should be for the removal of one of the standard. And the position of the operation is relatively high, which can lead to a large number of esophageal resection, and the length of esophageal resection is more than 3. The 5cm is sufficient. Therefore, how to implement a minimally invasive surgical approach to the upper and lower middle and upper mediastinal and abdominal lymph nodes is a hot research topic in the field of esophageal gastric junction adenocarcinoma.

Up to now, there is no reasonable standard minimally invasive surgery for treatment of type II esophageal gastric junction adenocarcinoma. The investigators sum up the experience of the past in the minimally invasive resection of esophageal cancer, and combine domestic and foreign research results. Pioneered by laparoscopic mobilization of the stomach and dissection of the abdominal field lymph node + thoracoscopic (left thoracic approach) to free the esophagus and cleaning + mirror under the purse string forceps esophagogastric aortic arch anastomosis under lower mediastinal lymph node, corresponding to the operation is the traditional through left thoracotomy combined with open operation on diaphragm. Can achieve the same with the traditional surgical resection of the tumor, while taking into account the characteristics of minimally invasive surgery. In this study, cases of type II esophageal gastric junction adenocarcinoma cases were collected from 120 patients with type II esophageal gastric junction adenocarcinoma by prospective randomized controlled clinical trial. Comparison of different surgical methods for patients with the safety of surgery, oncology resection range, the incidence of short-term complications. The effect of different surgical methods on the survival rate and quality of life of the two groups were compared with the postoperative follow-up. The surgical treatment of esophageal carcinoma with a reasonable level of type II type of esophageal gastric junction adenocarcinoma is improved, and the surgical treatment of esophageal gastric junction adenocarcinoma is improved.

ELIGIBILITY:
Can tolerate the cT1~3N0~1M0 phase II type II esophageal gastric junction adenocarcinoma patients with the corresponding operation, the past or present without radiotherapy, chemotherapy, nearly 5 years without any other malignant tumor history. According to the research design, random access to minimally invasive surgery group or traditional open surgery group. The follow-up procedure, if the cause of the disease or the treatment of the disease has been confirmed, such as the need for adjuvant chemotherapy, should be treated accordingly, according to the statistics appear to be accompanied by the interference to explain and deal with.

Inclusion Criteria:

A. under 70 years of age (taking into account the follow-up period); B. was performed in patients with cT1~3N0~1M0 type II type cTNM, C., F., D., e., and 5 years.

Exclusion Criteria:

I A., type III esophageal gastric junction adenocarcinoma; B. major organ function can not tolerate surgery; C. advanced patients.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the number of lymph nodes dissection | through study completion, an average of 1 year

SECONDARY OUTCOMES:
the number of positive lymph nodes | through study completion, an average of 1 year

OTHER OUTCOMES:
Bleeding volume in operation | through study completion, an average of 1 year
Operation time | through study completion, an average of 1 year
Postoperative hospitalization days | through study completion, an average of 1 year
Days after operation with thoracic drainage tube | through study completion, an average of 1 year
the volume of pleural fluid in the first 3 days after operation | through study completion, an average of 1 year
Hospitalization expenses | through study completion, an average of 1 year
Postoperative complications | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided